CLINICAL TRIAL: NCT04416373
Title: COVID-19 and Pregnancy Outcomes: a Portuguese Collaboration Study
Brief Title: COVID-19 and Pregnancy Outcomes
Acronym: COVID&PREG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidade Nova de Lisboa (Other)
Responsible Party: Sponsor
Other Study IDs: COVID&PREG
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Coronavirus Infection; Pregnancy Complications; Vertical Transmission of Infectious Disease; Breastfeeding; Neonatal Infection
MeSH Terms: conditions — Coronavirus Infections; Pregnancy Complications; Breast Feeding | interventions — COVID-19 Nucleic Acid Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: RT PCR SARS-CoV-2 — Positive SARS-CoV-2 RT PCR in nasopharyngeal/oral swab tests or presence of IgM in blood samples
  Other Names: SARS-COV-2 Serologic test

SUMMARY:
This is a multicenter prospective study that aims to investigate the clinical impact of SARS-CoV-2 infection in pregnant women, pregnancy outcomes and perinatal transmission.

DETAILED DESCRIPTION:
This is a cohort study of pregnant women confirmed positive for SARS-CoV-2 infection. Data will be collected in Portuguese maternities that agreed to collaborate in this study.

Pregnant women are tested during hospital admission by using nasopharyngeal/oral swabs for SARS-CoV-2 RT PCR as part of a universal testing policy. Maternal demographic data (age, comorbidities, parity, smoking habits), COVID-19 related data (symptoms, diagnostic tests, therapy used and ICU admission), gestational age at SARS-CoV-2 confirmed infection, pregnancy outcomes (gestational complications, gestational age at birth, mode of delivery) and neonatal outcome (birthweight and Apgar score, RT PCR neonate results) and breastfeeding strategies will be evaluated.

ELIGIBILITY:
Inclusion Criteria: Pregnant women infected with Sars-Cov-2. Delivery at Portuguese maternities.

Exclusion Criteria: RT PCR SARS-CoV-2 negative.

-

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pregnant women infected with Sars-Cov-2 from 6 to 41 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-03-22 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 Neonatal Infection | 7 days
  Positive Sars-Cov-2 RT PCR in nasopharyngeal/oral swab tests or presence of IgM in blood samples

SECONDARY OUTCOMES:
Perinatal mortality | 35 weeks
  stillbirths and deaths in the first week of life
ICU maternal admission | 35 weeks
  maternal ICU admission due to COVID-19
5 minute Apgar Score < 7 | 1 day
  Newborn 5 minute Apgar Score < 7
Preterm labour | 35 weeks
  Delivery between 24 and 36 weeks
PPROM | 35 weeks
  Preterm premature rupture of the membranes between 24 and 36 weeks
Miscarriage | 14 weeks
  spontaneous pregnancy loss before 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Medical School - UNL, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Undecided